CLINICAL TRIAL: NCT05198024
Title: Effects of Nutrition Education in Cardiac Rehabilitation Patients; a 3-arm Randomized Controlled Trial
Brief Title: Nutrition Education in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Sinclair (Other)
Responsible Party: Sponsor-Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Organization: University of Central Lancashire (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nutrition Education
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Placebo Comparator): Where patients access to two exercise classes per week and all facilities as part of their cardiac rehabilitation. In addition to this, patients in this group took part in the 'Biggest loser' program in which the patients attended weekly sessions outside of their usual exercise class times. Each session follows a specific theme based on British Heart Foundation healthy eating guidelines.
  Participants will undergo this approach for 6-weeks and then switch to usual care for 6-weeks.
  Interventions: Behavioral: Nutrition knowledge
- Usual care plus biggest loser (Experimental): Where patients access to two exercise classes per week and all facilities as part of their cardiac rehabilitation. In addition to this, patients in this group took part in the 'Biggest loser' program in which the patients attended weekly sessions outside of their usual exercise class times. Each session follows a specific theme based on British Heart Foundation healthy eating guidelines.
  Participants will undergo this approach for 6-weeks and then switch to usual care for 6-weeks.
  Interventions: Behavioral: Nutrition knowledge
- Usual care plus new education programme (Experimental): Where patients access to two exercise classes per week and all facilities as part of their cardiac rehabilitation. In addition to this, patients in this group too part in a new education programme (anecdotally referred to as "Healthy Heart Happy You") in which the same weekly topics as the biggest loser are covered yet with bespoke information regarding portion sizes and recipes provided each week and patients given a challenge each week in relation to the topic being covered e.g. include more vegetables.
  Participants will undergo this approach for 6-weeks and then switch to usual care for 6-weeks.
  Interventions: Behavioral: Nutrition knowledge

INTERVENTIONS:
Behavioral: Nutrition knowledge — Nutrition knowledge either 'Usual care plus new education programme' or 'Usual care plus biggest loser'

SUMMARY:
Coronary heart disease is one of the United Kingdom's biggest killers. In the UK alone 175,000 myocardial infarctions are recorded annually. To lower the financial burden on the National Health Service, cardiac rehabilitation facilitates a systematic and multidisciplinary approach to secondary prevention aimed to improve functional capacity and health-related quality of life, lower rehospitalisation rates and reduce all-cause and cardiovascular mortality with exercise training being the cornerstones. The effectiveness of

Cardiac rehabilitation programmes in delivering effective secondary prevention has long been established. Improvements are recorded in cardiovascular endurance, muscular strength and endurance, balance, co-ordination, and quality of life. However, many patients see little or no change in body mass and body mass index, an independent risk factor for coronary heart disease. Interestingly, the inclusion of nutrition education is rarely reported within specific Cardiac rehabilitation settings, therefore evidence of best practice remains elusive and warrants further investigation.

The aim of this trial is to compare:

* Usual care - Where patients access to two exercise classes per week and all facilities normally available as part of their cardiac rehabilitation programme. Patients in this group will undergo this approach for 12-weeks.
* Usual care + Biggest loser - In addition to Usual care, patients in this group took part in the 'Biggest loser' program in which the patients attended weekly sessions outside of their usual exercise class times. Each session follows a specific theme based on British Heart Foundation healthy eating guidelines. Participants will undergo this approach for 6-weeks and then switch to usual care for 6-weeks.
* Usual care + New Education programme. In addition to Usual care, the same weekly topics as the biggest loser are covered yet with bespoke information regarding portion sizes and recipes provided each week and patients given a challenge each week in relation to the topic being covered e.g. include more vegetables. Participants will undergo this approach for 6-weeks and then switch to usual care for 6-weeks.

Patients will be tested at baseline, 6-weeks and 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Engaged in phase IV cardiac rehabilitation program
* Patient has read and understood the Patient Information Sheet
* Clinically stable (symptoms and medication)

Exclusion Criteria:

* Clinically Unstable (symptoms and medication)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor
Blood pressure | 6-weeks
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor
Blood pressure | 12-weeks
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 6-weeks
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 12-weeks
  Ratio of waist to hip circumference - measured using anthropocentric tape
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 6-weeks
  Capillary blood glucose - mmol/L
Blood glucose | 12-weeks
  Capillary blood glucose - mmol/L
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 6-weeks
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 12-weeks
  Capillary blood triglycerides - mmol/L
Blood cholesterol | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol | 6-weeks
  Capillary blood cholesterol - mmol/L
Blood cholesterol | 12-weeks
  Capillary blood cholesterol - mmol/L
Body mass | Baseline
  Body mass (kg)
Body mass | 6-weeks
  Body mass (kg)
Body mass | 12-weeks
  Body mass (kg)
Body mass index | Baseline
  Body mass index kg/m2
Body mass index | 6-weeks
  Body mass index kg/m2
Body mass index | 12-weeks
  Body mass index kg/m2
Waist circumference | Baseline
  Waist circumference (cm)
Waist circumference | 6-weeks
  Waist circumference (cm)
Waist circumference | 12-weeks
  Waist circumference (cm)
Mediterranean Diet score | Baseline
  Mediterranean score obtained from the Mediterranean Diet Assessment tool. A lower score means higher risk from cardiovascular disease. The scale has a score range from 0-14.
Mediterranean Diet score | 6-weeks
  Mediterranean score obtained from the Mediterranean Diet Assessment tool. A lower score means higher risk from cardiovascular disease. The scale has a score range from 0-14.
Mediterranean Diet score | 12-weeks
  Mediterranean score obtained from the Mediterranean Diet Assessment tool. A lower score means higher risk from cardiovascular disease. The scale has a score range from 0-14.
Total energy | Baseline
  Total daily energy (kcal) taken from a 4-day diet diary
Total energy | 6-weeks
  Total daily energy (kcal) taken from a 4-day diet diary
Total energy | 12-weeks
  Total daily energy (kcal) taken from a 4-day diet diary
Calcium intake | Baseline
  Calcium intake per day (mg/day) taken from a 4-day diet diary
Calcium intake | 6-weeks
  Calcium intake per day (mg/day) taken from a 4-day diet diary
Calcium intake | 12-weeks
  Calcium intake per day (mg/day) taken from a 4-day diet diary
Vitamin B12 intake | Baseline
  Vitamin B12 (ug) intake per day taken from a 4-day diet diary
Vitamin B12 intake | 6-weeks
  Vitamin B12 (ug) intake per day taken from a 4-day diet diary
Vitamin B12 intake | 12-weeks
  Vitamin B12 (ug) intake per day taken from a 4-day diet diary
Vitamin B6 intake | Baseline
  Vitamin B6 (mg) intake per day taken from a 4-day diet diary
Vitamin B6 intake | 6-weeks
  Vitamin B6 (mg) intake per day taken from a 4-day diet diary
Vitamin B6 intake | 12-weeks
  Vitamin B6 (mg) intake per day taken from a 4-day diet diary
Folate intake | Baseline
  Folate (ug) intake per day taken from a 4-day diet diary
Folate intake | 6-weeks
  Folate (ug) intake per day taken from a 4-day diet diary
Folate intake | 12-weeks
  Folate (ug) intake per day taken from a 4-day diet diary
Vitamin A intake | Baseline
  Vitamin A (ug) intake per day taken from a 4-day diet diary
Vitamin A intake | 6-weeks
  Vitamin A (ug) intake per day taken from a 4-day diet diary
Vitamin A intake | 12-weeks
  Vitamin A (ug) intake per day taken from a 4-day diet diary
Vitamin C intake | Baseline
  Vitamin C (mg) intake per day taken from a 4-day diet diary
Vitamin C intake | 6-weeks
  Vitamin C (mg) intake per day taken from a 4-day diet diary
Vitamin C intake | 12-weeks
  Vitamin C (mg) intake per day taken from a 4-day diet diary
Vitamin D intake | Baseline
  Vitamin D (ug) intake per day taken from a 4-day diet diary
Vitamin D intake | 6-weeks
  Vitamin D (ug) intake per day taken from a 4-day diet diary
Vitamin D intake | 12-weeks
  Vitamin D (ug) intake per day taken from a 4-day diet diary
Vitamin E intake | Baseline
  Vitamin E (mg) intake per day taken from a 4-day diet diary
Vitamin E intake | 6-weeks
  Vitamin E (mg) intake per day taken from a 4-day diet diary
Vitamin E intake | 12-weeks
  Vitamin E (mg) intake per day taken from a 4-day diet diary
Thiamine intake | Baseline
  Thiamine (mg) intake per day taken from a 4-day diet diary
Thiamine intake | 6-weeks
  Thiamine (mg) intake per day taken from a 4-day diet diary
Thiamine intake | 12-weeks
  Thiamine (mg) intake per day taken from a 4-day diet diary
Riboflavin intake | Baseline
  Riboflavin (mg) intake per day taken from a 4-day diet diary
Riboflavin intake | 6-weeks
  Riboflavin (mg) intake per day taken from a 4-day diet diary
Riboflavin intake | 12-weeks
  Riboflavin (mg) intake per day taken from a 4-day diet diary
Selenium intake | Baseline
  Selenium (ug) intake per day taken from a 4-day diet diary
Selenium intake | 6-weeks
  Selenium (ug) intake per day taken from a 4-day diet diary
Selenium intake | 12-weeks
  Selenium (ug) intake per day taken from a 4-day diet diary
Zinc intake | Baseline
  Zinc (mg) intake per day taken from a 4-day diet diary
Zinc intake | 6-weeks
  Zinc (mg) intake per day taken from a 4-day diet diary
Zinc intake | 12-weeks
  Zinc (mg) intake per day taken from a 4-day diet diary
Sodium intake | Baseline
  Sodium (mg) intake per day taken from a 4-day diet diary
Sodium intake | 6-weeks
  Sodium (mg) intake per day taken from a 4-day diet diary
Sodium intake | 12-weeks
  Sodium (mg) intake per day taken from a 4-day diet diary
Carbohydrate intake | Baseline
  Carbohydrate (g) intake per day taken from a 4-day diet diary
Carbohydrate intake | 6-weeks
  Carbohydrate (g) intake per day taken from a 4-day diet diary
Carbohydrate intake | 12-weeks
  Carbohydrate (g) intake per day taken from a 4-day diet diary
Fat intake | Baseline
  Fat (g) intake per day taken from a 4-day diet diary
Fat intake | 6-weeks
  Fat (g) intake per day taken from a 4-day diet diary
Fat intake | 12-weeks
  Fat (g) intake per day taken from a 4-day diet diary
Sugar intake | Baseline
  Sugar (g) intake per day taken from a 4-day diet diary
Sugar intake | 6-weeks
  Sugar (g) intake per day taken from a 4-day diet diary
Sugar intake | 12-weeks
  Sugar (g) intake per day taken from a 4-day diet diary
Fibre intake | Baseline
  Fibre (g) intake per day taken from a 4-day diet diary
Fibre intake | 6-weeks
  Fibre (g) intake per day taken from a 4-day diet diary
Fibre intake | 12-weeks
  Fibre (g) intake per day taken from a 4-day diet diary
Starch intake | Baseline
  Starch (g) intake per day taken from a 4-day diet diary
Starch intake | 6-weeks
  Starch (g) intake per day taken from a 4-day diet diary
Starch intake | 12-weeks
  Starch (g) intake per day taken from a 4-day diet diary
Protein intake | Baseline
  Protein (g) intake per day taken from a 4-day diet diary
Protein intake | 6-weeks
  Protein (g) intake per day taken from a 4-day diet diary
Protein intake | 12-weeks
  Protein (g) intake per day taken from a 4-day diet diary
Saturated fat intake | Baseline
  Saturated fat (g) intake per day taken from a 4-day diet diary
Saturated fat intake | 6-weeks
  Saturated fat (g) intake per day taken from a 4-day diet diary
Saturated fat intake | 12-weeks
  Saturated fat (g) intake per day taken from a 4-day diet diary
Monounsaturated fat intake | Baseline
  Monounsaturated fat (g) intake per day taken from a 4-day diet diary
Monounsaturated fat intake | 6-weeks
  Monounsaturated fat (g) intake per day taken from a 4-day diet diary
Monounsaturated fat intake | 12-weeks
  Monounsaturated fat (g) intake per day taken from a 4-day diet diary
Polyunsaturated fat intake | Baseline
  Polyunsaturated fat (g) intake per day taken from a 4-day diet diary
Polyunsaturated fat intake | 6-weeks
  Polyunsaturated fat (g) intake per day taken from a 4-day diet diary
Polyunsaturated fat intake | 12-weeks
  Polyunsaturated fat (g) intake per day taken from a 4-day diet diary

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom